CLINICAL TRIAL: NCT06118190
Title: The Effectiveness of Mesotherapy (Lidocaine and Proxicam) in the Treatment of Chronic Migraine
Brief Title: Mesotherapy in the Treatment of Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Elif Ozyigit, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KAEK/2022.11.225
Record Dates: First submitted 2023-10-30; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Chronic Migraine, Headache
Keywords: Mesotherapy; Chronic Migraine; pain; muscle; headache
MeSH Terms: conditions — Headache; Pain

STUDY DESIGN:
Intervention Model Description: Retrospective analysis of the group that received treatment
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mesotherapy (Experimental): All participants who received mesotherapy were monitored regularly for the following three months to assess their prognosis and ensure patient adherence to treatment.
  Interventions: Drug: Lidocain

INTERVENTIONS:
Drug: Lidocain — All participants treated with procaine and lidocaine injection for treatment.
  Other Names: Proxicam

SUMMARY:
Mesotherapy is a type of injection frequently used in clinics. It is a treatment procedure that involves the injection of some drugs under the skin or into the skin. Mesotherapy is used in musculoskeletal system diseases, but it is reported that the effects of its use in migraine are uncertain.

DETAILED DESCRIPTION:
Migraine is one of the types of headaches. For the diagnosis of chronic migraine, the headache must last more than 15 days. Nerve blocks, oral medication and neuromodulation are recommended for migraine treatment.Mesotherapy is a type of injection frequently used in clinics. It is a treatment procedure that involves the injection of some drugs under the skin or into the skin. Mesotherapy is used in musculoskeletal system diseases, but it is reported that the effects of its use in migraine are uncertain. This study was planned to show the effectiveness of mesotherapy in patients with migraine.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of chronic migraine disease

Exclusion Criteria:

* Infection disease
* Thyroid disease
* Anemia disease
* Systemic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2023-10-29 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline
  VAS rates pain on a scale of zero to 10. It is explained to the participant that 10 points means unbearable pain, zero points means no pain, and the patient is asked to rate his pain between zero and ten. Higher scores indicate increased pain severity
Visual Analog Scale (VAS) | 4th week
  VAS rates pain on a scale of zero to 10. It is explained to the participant that 10 points means unbearable pain, zero points means no pain, and the patient is asked to rate his pain between zero and ten. Higher scores indicate increased pain severity
Visual Analog Scale (VAS) | 8th week
  VAS rates pain on a scale of zero to 10. It is explained to the participant that 10 points means unbearable pain, zero points means no pain, and the patient is asked to rate his pain between zero and ten. Higher scores indicate increased pain severity
Visual Analog Scale (VAS) | 12 th week
  VAS rates pain on a scale of zero to 10. It is explained to the participant that 10 points means unbearable pain, zero points means no pain, and the patient is asked to rate his pain between zero and ten. Higher scores indicate increased pain severity
The frequency of painful days per month | Baseline
  The participant is asked how many days she/he feels pain in a month.Higher numbers indicate increased frequency of painful days
The frequency of painful days per month | 4th week
  The participant is asked how many days she/he feels pain in a month.Higher numbers indicate increased frequency of painful days
The frequency of painful days per month | 8th week
  The participant is asked how many days she/he feels pain in a month.Higher numbers indicate increased frequency of painful days
The frequency of painful days per month | 12th week
  The participant is asked how many days she/he feels pain in a month.Higher numbers indicate increased frequency of painful days

SECONDARY OUTCOMES:
Duration of attack per month | Baseline
  The participant is questioned about how long each attack lasts within a month. Increased periods indicate prolonged symptom duration.
Duration of attack per month | 4th week
  The participant is questioned about how long each attack lasts within a month. Increased periods indicate prolonged symptom duration.
Duration of attack per month | 8th week
  The participant is questioned about how long each attack lasts within a month. Increased periods indicate prolonged symptom duration.
Duration of attack per month | 12th week
  The participant is questioned about how long each attack lasts within a month. Increased periods indicate prolonged symptom duration.
the number of analgesic per month | Baseline
  The participant is asked how many times he/she uses analgesic medication in a month. Higher numbers indicate an increased need for medical treatment
the number of analgesic per month | 4th week
  The participant is asked how many times he/she uses analgesic medication in a month. Higher numbers indicate an increased need for medical treatment
the number of analgesic per month | 8th week
  The participant is asked how many times he/she uses analgesic medication in a month. Higher numbers indicate an increased need for medical treatment
the number of analgesic per month | 12th week
  The participant is asked how many times he/she uses analgesic medication in a month. Higher numbers indicate an increased need for medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elif Ozyigit, MD, Principal Investigator — Kanuni Sultan Suleyman Research and Training Hospital
Locations (1):
- Kanni Sultan Suleyman Research and Training Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The investigators were undecided

REFERENCES:
- [Background] Costantino C, Marangio E, Coruzzi G. Mesotherapy versus Systemic Therapy in the Treatment of Acute Low Back Pain: A Randomized Trial. Evid Based Complement Alternat Med. 2011;2011:317183. doi: 10.1155/2011/317183. Epub 2010 Sep 1. PMID 20953425
- [Background] Ravishankar K, Tayade H, Mandlik R. Sublingual piroxicam in migraine without aura. J Assoc Physicians India. 2011 Aug;59:494-7. PMID 21887905